CLINICAL TRIAL: NCT06758752
Title: Evaluation of Therapeutic Effects of ZAX.1400.EC.02 a Herbal Compound on Clinical Signs of Skin in Eczema Patients
Brief Title: A Herbal Compound for Eczema
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fasa University of Medical Sciences (Other)
Collaborators: Herbmedx Co (Industry); Zarrin Avaye Kowsar Salamat (ZAX company) (Unknown)
Responsible Party: Principal Investigator, Akbar Farjadfar, Principle-Investigator, Fasa University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRCT20210218050404N3
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-09

CONDITIONS: Eczema; Atopic Dermatitis; Inflammation
Keywords: Eczema; Atopic Dermatitis; Inflammation; Anti-inflammatory; Herbal medicines; Natural Products
MeSH Terms: conditions — Eczema; Dermatitis, Atopic; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical ZAX.1400.EC.02 (Experimental): ZAX.1400.EC.02, applied topically twice daily for 3 weeks after enrolment
  Interventions: Dietary Supplement: ZAX.1400.EC.02
- Placebo (Placebo Comparator): Placebo, applied topically twice daily for 3 weeks after enrolment
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: ZAX.1400.EC.02 — ZAX.1400.EC.02, applied twice daily for 3 weeks after enrolment
  Arms: Topical ZAX.1400.EC.02
Drug: Placebo — Placebo, applied twice daily for 3 weeks after enrolment
  Arms: Placebo

SUMMARY:
The goal of this interventional clinical trial study is to compare ZAX.1400.EC.02 and placebo in Eczema patients. The main question it aims to answer is:

• Can treatment with ZAX.1400.EC.02 for 3 weeks improve clinical signs of skin in Eczema patients? Participants will be divided into two groups. One group will use ZAX.1400.EC.02 topically twice daily for 3 weeks and the other group will use placebo topically twice daily for 3 weeks.

Researchers will compare treatment and placebo groups to see if there is any improvement in the clinical signs of skin caused by Eczema after treatment with ZAX.1400.EC.02 for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of the disease by a doctor
* Age range between 18 and 60 years
* Both sexes (male and female)
* Having written informed consent to participate in the study
* Lack of allergy to food and health products
* Absence of underlying diseases and immune deficiency
* Absence of pregnancy and breastfeeding
* Absence of blisters and infection caused by the disease

Exclusion Criteria:

* Non-consent of the doctor directly responsible for the patient
* Incidence of drug product allergy
* Occurrence of symptoms of skin, digestive, liver or kidney diseases
* Patients lack of consent to continue for any reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Dermatology Life Quality Index (DLQI) score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  DLQI score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42

SECONDARY OUTCOMES:
Change From Baseline in Percent Body Surface Area (%BSA) at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Body Surface Area (BSA) is a numerical score used to measure the physician's assessment of the percentage of the participant's total BSA involved with psoriasis. BSA = SQRT ((height (cm) X weight (kg))/3600) BSA is in m2, W is weight in kg, and H is height in cm. Total body Surface Area (BSA) in meters squared %Body Surface Area Affected the "Rule of Nine" was be used
Change From Baseline in erythema score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Erythema score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in Swelling score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Swelling score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in pruritus score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Pruritus score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in flake score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Flake score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin dryness score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin dryness score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin irritation score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin irritation score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in pain score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Pain score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin scratch score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin scratch score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin scar score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin scar score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin thickness score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin thickness score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42
Change From Baseline in skin rashes score at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42 | Baseline and Weeks 1, 2, 3, 4, 5, and 6
  Skin rashes score will be assessed at Day0 (Baseline), Day7, Day14, Day21, Day28, Day35, and Day42

CONTACTS AND LOCATIONS:
Locations (1):
- Fasa university of medical sciences, Fasa, Fars, Iran